CLINICAL TRIAL: NCT04726696
Title: Clarification of Nurses' Expected Role in Health Promotion: Study Protocol of an Exploratory Clustered Randomised Controlled Trial for the ROLE-AP Program
Brief Title: Clarification of Nurses' Expected Role in Health Promotion
Acronym: ROLE-AP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Gobierno de Navarra (Unknown); Universidad Pública de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GºNa15/19
Record Dates: First submitted 2021-01-14; First posted 2021-01-27 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2020-07

CONDITIONS: Role, Nurses
Keywords: Role clarification; Nurses' role; Health promotion; Prevention

STUDY DESIGN:
Intervention Model Description: The study will be conducted in the province of Navarra (Spain), in the primary health care service. The study will follow a cluster randomised design with primary care teams (PCT) as sampling units. A PCT consists of a group of family physicians who work in close cooperation with nurses and social workers to offer primary care services to registered individuals in the area. Each cluster will be randomly assigned to one of the two groups, control or intervention. The main reason for using a cluster design is to avoid contamination, which could occur among nurses working in the same PCT. This is more likely given the particular characteristics of this complex intervention in which masking is not possible. The R software (version 3.3.0) will be used to choose an allocation at random. The randomisation of the study groups will be stratified according to the scope of work (rural / urban), to guarantee the representativeness of the different segments of the study population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): None intervention to be administered, they continue their normal routine.
- Intervention group (Experimental): ROLE-AP is a multifaceted program offered over a month period to participating primary care nurses and includes three interactive workshops. Each workshop will be 4 hours long.
  Interventions: Behavioral: ROLE-AP programme

INTERVENTIONS:
Behavioral: ROLE-AP programme — The intervention group will be split in two groups of 7-8 primary care nurses each. These two groups will receive the ROLE-AP program over a three weeks period. Each workshop will be divided into two sessions of 90-120min. The first workshop focuses on the clarification of health promotion concepts and the discussion of the state of nursing practice in health promotion. Participants will discuss the misalignments between this description of nursing practice and the ideal one portrayed by the Ottawa Charter. The second workshop will allow the presentation of the objectives of the health care organization, showing its alignment with the Ottawa Charter areas of action. In addition, it will present a standardized instrument that reflects expectations about nurses' activities in health promotion that will serve for discussing and realigning participants' expectations on nurses' role in health promotion. The third workshop will continue with the discussion of nurses' expected activities.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to implement and evaluate ROLE-AP, a multi-component program to clarify primary care nurses' expected role in health promotion. It is hypothesized that, in comparison with the control group, participants in the experimental group will increase their degree of agreement on nurses' role in health promotion.

DETAILED DESCRIPTION:
Role confusion is hampering the development of primary care nurses' capacity for health promotion. Organizations can implement role clarification programs to develop the description of an expected role in the organization and reduce the negative effects of role confusion. Literature on role clarification interventions reveal that they are complex interventions seeking discussion to reach agreement between professionals about the expected role activities. However, such interventions have shown several methodological shortcomings. This study aims to implement and evaluate a multi-component program to clarify primary care nurses' role in health promotion. An exploratory clinical trial will help evaluate the preliminary efficacy and understand if an intervention of these characteristics is feasible, if its components are appropriate and / or if it is accepted by the participants. This is a pilot cluster randomized exploratory trial, which corresponds to Phase II of the Medical Research Council (MRC) framework for the development and evaluation of clinical trials in complex interventions. The study will be conducted in the province of Navarra (Spain), in the primary health care service. The study will follow a cluster randomised design with primary care teams (PCT) as sampling units. A PCT consists of a group of family physicians who work in close cooperation with nurses and social workers to offer primary care services to registered individuals in the area. Each cluster will be randomly assigned to one of the two groups, control or intervention. The main reason for using a cluster design is to avoid contamination, which could occur among nurses working in the same PCT. The randomisation of the study groups will be stratified according to the scope of work (rural / urban), to guarantee the representativeness of the different segments of the study population. It has been considered that nurses' activities and the perception they may have about their health promoting role may be conditioned by two factors: the organization and structure of the PCT and the characteristics of the populations they attend. These two factors may vary depending on the team attending rural or urban population, so it will be considered as a possible confusing variable. The control group will continue with their routine.

ELIGIBILITY:
Inclusion Criteria:

* being a primary care nurse in the Navarre health service.
* have two years of professional experience in primary health care
* be a nurse attending either adult or pediatric population
* have signed the consent form for participation in the study

Exclusion Criteria:

- not planning to be in clinical practice for the whole duration of the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-21 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes on nurses' agreement on their role using the Spanish version of "Nurses' Role in Health Promotion Questionnaire" | Baseline (T0), immediately after intervention (T1) and 3 months follow up (T2)
  Nurses will complete the questionnaire at 3 time points.

OTHER OUTCOMES:
Barriers to program implementation assessed by the researcher's field diary (Feasibility) | Baseline (T0)
  Explored by the researchers' field diary, without using any scale. It will collect qualitative data related to barriers/facilitators to the randomization and recruitment process, degree of collaboration of the primary care managers, resources and materials used and characteristics of the context in which the intervention takes place.
Fidelity of the program assessed by the "ROLE-AP program checklist" (Quality) | During the intervention
  Fidelity will be evaluated through structured observations of each program session. The checklist will contain the following information: compliance with the programmed activities, order of activities and time spent for each activity.
Acceptability of the program by nurses, assessed by the "Nurses' satisfaction with the ROLE-AP program questionnaire" | Immediately after intervention
  The acceptance and satisfaction of the participants with the program will be measured through a questionnaire prepared for this purpose. Three closed questions will assess the degree of satisfaction with the program, the recommendation and need for programs of these characteristics.
Quality of the program assessed by the "Nurses' satisfaction with the ROLE-AP program questionnaire" and debriefing sessions. | During the intervention and Immediately after intervention
  The questionnaire contains three open questions to know nurses' opinions about the materials used, the role of the facilitator and possible suggestions for the improvement of the program.
  The debriefing sessions will take place after each session of the program. The script will contain questions about positive and negative aspects of the program perceived by the research team.
Effect size assessed by the Cohen's formula | Immediately after intervention
  The Cohen's formula will be used to estimate the size effect for a definitive randomized clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Iriarte, Principal Investigator — University of Navarra
Locations (1):
- University of Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Derived] Iriarte-Roteta A, Lopez-Dicastillo O, Mujika A, Antonanzas-Baztan E, Hernantes N, Galan Espinilla MJ, Pumar-Mendez MJ. Building capacity for health promotion by addressing nurses' role confusion: Study protocol of a pilot clustered randomised controlled trial. J Adv Nurs. 2021 Nov;77(11):4574-4585. doi: 10.1111/jan.15018. Epub 2021 Aug 21. PMID 34418139